CLINICAL TRIAL: NCT00349037
Title: A Prospective, Randomised, Double Blind, Placebo-Controlled Study to Assess the Efficacy of a Trivalent (A/New Caledonia/20/99, A/Panama/2007/99, B/Jiangsu/10/20) DNA Influenza Vaccine Administered by Particle Mediated Epidermal Delivery (PMED) Against a Controlled Influenza Virus Challenge.
Brief Title: Study of the Ability of a Flu Vaccine to Prevent Flu Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PowderMed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PM FLS-002
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Influenza
Keywords: DNA vaccine; influenza; immunogenicity; tolerability; PMED; efficacy; challenge virus
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Trivalent DNA vaccine with and without pPJV2012 administered by PMED

SUMMARY:
The purpose of this study is to evaluate how effective the vaccine is at preventing subjects developing flu symptoms after they are directly exposed to flu virus. The study will also evaluate how well the vaccine is tolerated at sites where administrations are given, any effects it may have on subjects' wellbeing and whether it can produce antibody responses in the body

DETAILED DESCRIPTION:
Influenza is a contagious disease of the upper airways and the lungs. It rapidly spreads around the world in seasonal epidemics, killing hundreds of thousands of people and having high economic consequences due to healthcare costs and lost productivity. Each year governments recommend groups who are at risk of influenza or its complications to receive influenza vaccination. Current vaccine supply is not sufficient to meet the demand if this recommendation were to be taken up by all. This study will evaluate PowderMed's Particle Mediated Epidermal Delivery (PMED) DNA vaccine for influenza as a potential alternative to existing vaccine technologies. This study will assess how effective two different PMED vaccine combinations are at preventing subjects developing influenza following exposure to flu virus 56 days after a single dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult volunteers (women must be of non child-bearing potential)

Provided written informed consent

Exclusion Criteria:

No significant concomitant illness

No allergy to gold

No immunosuppression due to disease or treatment

Pre-existing protective level of antibody against the challenge virus strain

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105
Dates: Start 2006-09; Study Completion 2007-01

PRIMARY OUTCOMES:
Efficacy of the vaccine in preventing symptoms of influenza-like illness

SECONDARY OUTCOMES:
Safety and tolerability - AEs and laboratory tests. Immunogenicity of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mant, BSc, FRCP, FFPM, Principal Investigator — GDRU
Locations (1):
- GDRU Quintiles Ltd, London, United Kingdom